CLINICAL TRIAL: NCT03582501
Title: Physiology of the Early Stage of Hemorrhage and Early Identification of Progression Toward Hemodynamic Instability in Humans for Validation of Current Machine Learning Models
Brief Title: Measurement of Hemodynamic Responses to Lower Body Negative Pressure
Acronym: LBNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Timothy B. Curry, Vice Chair, Dept of Anesthesiology and Perioperative Medicine, Primary Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-002695
Record Dates: First submitted 2018-06-26; First posted 2018-07-11 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Hypotension and Shock
MeSH Terms: conditions — Hypotension; Shock | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): All volunteers will be studied at rest and during experimental condition (lower body negative pressure)
  Interventions: Other: Lower body negative pressure

INTERVENTIONS:
Other: Lower body negative pressure — Simulated hypovolemia by applied suction to lower extremities to cause venous pooling.

SUMMARY:
This study will be collecting data on participants undergoing lower body negative pressure (LBNP) to simulate progressive blood loss. The goal of the study is to collect data to allow for development of an algorithm with machine learning to predict blood pressure responses to hypovolemia by analyzing the arterial waveforms collected during LBNP.

DETAILED DESCRIPTION:
Death from exsanguination continues to be a major problem in combat casualty care and the care of civilians subjected to trauma. The ability to detect significant blood loss using traditional vital signs (heart rate, blood pressure) is marginal due to a variety of compensatory mechanisms that maintain blood pressure in the face of marked reductions in circulating blood volume. Along these lines, it is critical to develop monitoring devices and algorithms to non-invasively assess central blood volume in humans for the purposes of facilitating more timely interventions. The standard way to simulate hemorrhage in humans is to use Lower Body Negative Pressure (LBNP). In this technique, the lower body of a supine volunteer is enclosed in an airtight container while suction is applied to cause venous pooling in the legs and reduce central blood volume. This technique generates many physiological adaptations that are similar to that observed during blood loss studies in animals and human volunteers. Thus, the purpose of this study is to obtain data for use in developing monitoring technology to detect hemorrhage and other surrogate markers of central blood volume in humans.

ELIGIBILITY:
Inclusion criteria:

18-55 year of age Non-smoker No history of hypertension No history of diabetes No history of coronary artery disease No history of neurologic disease

Exclusion criteria Prescribed medications other than birth control Inability to lie flat for two hours BMI > 30 kg/m2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Blood pressure | One day of study visit
  Arterial blood pressure prior to and during lower body negative pressure

SECONDARY OUTCOMES:
Heart rate | One day of study visit
  Heart rate prior to and during lower body negative pressure

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Curry, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota